CLINICAL TRIAL: NCT02691494
Title: A Phase 3 Study to Evaluate the Efficacy and Safety of Elagolix in Combination With Estradiol/Norethindrone Acetate for the Management of Heavy Menstrual Bleeding Associated With Uterine Fibroids in Premenopausal Women
Brief Title: Efficacy and Safety of Elagolix in Combination With Estradiol/Norethindrone Acetate for the Management of Heavy Menstrual Bleeding Associated With Uterine Fibroids in Premenopausal Women (Replicate Study)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M12-817
Record Dates: First submitted 2016-02-22; First posted 2016-02-25 (Estimated); Results first posted 2020-06-30 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Uterine Fibroids; Heavy Menstrual Bleeding
Keywords: Elagolix; Elagolix Sodium; Heavy uterine bleeding; Heavy menstrual bleeding (HMB); Leiomyomata; Menorrhagia; ABT-620; Elagolix + E2/NETA (Elagolix + Norethindrone acetate)
MeSH Terms: conditions — Leiomyoma; Menorrhagia | interventions — elagolix; Estradiol; Norethindrone Acetate; estradiol, norethindrone drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo for both elagolix twice daily (BID) and norethindrone acetate (E2/ NETA) once daily (QD)
  Interventions: Drug: Placebo for Estradiol/Norethindrone Acetate; Drug: Placebo for Elagolix
- Elagolix (Experimental): Elagolix 300 mg BID and placebo for E2/NETA (estradiol 1.0 mg/norethindrone acetate 0.5 mg) QD
  Interventions: Drug: Elagolix; Drug: Placebo for Estradiol/Norethindrone Acetate
- Elagolix + E2/NETA (Experimental): Elagolix 300 mg BID and E2/NETA (estradiol 1.0 mg/norethindrone acetate 0.5 mg) QD
  Interventions: Drug: Elagolix; Drug: Estradiol/Norethindrone Acetate

INTERVENTIONS:
Drug: Elagolix — Film-coated tablets
  Other Names: ABT-620; elagolix sodium
  Arms: Elagolix; Elagolix + E2/NETA
Drug: Placebo for Estradiol/Norethindrone Acetate — Placebo capsules
  Arms: Elagolix; Placebo
Drug: Estradiol/Norethindrone Acetate — Commercially-available E2/NETA tablets were over-encapsulated to maintain study blinding.
  Other Names: E2/NETA
  Arms: Elagolix + E2/NETA
Drug: Placebo for Elagolix — Film-coated placebo tablets
  Arms: Placebo

SUMMARY:
This study seeks to evaluate the efficacy, safety and tolerability of elagolix alone and in combination with estradiol/norethindrone acetate for the management of heavy menstrual bleeding associated with uterine fibroids in premenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a premenopausal female at the time of Screening.
* Subject has a diagnosis of uterine fibroids documented by a pelvic ultrasound (transabdominal ultrasound/transvaginal ultrasound).
* Subject has heavy menstrual bleeding associated with uterine fibroids as evidenced by menstrual blood loss > 80 mL during each of two screening menses as measured by the alkaline hematin method.
* Subject has negative urine and/or serum pregnancy test in Screening and just prior to first dose.
* Subject has an adequate endometrial biopsy performed during Screening, the results of which show no clinically significant endometrial pathology.

Exclusion Criteria:

* Subject has screening pelvic ultrasound or saline infusion sonohysterography results that show a clinically significant gynecological disorder.
* Subject has history of osteoporosis or other metabolic bone disease.
* Subject has clinically significant abnormalities in clinical chemistry, hematology, or urinalysis.
* Subject has a history of major depression or post-traumatic stress disorder (PTSD) within 2 years of screening, OR a history of other major psychiatric disorder at any time (e.g., schizophrenia, bipolar disorder).
* Subject is using any systemic corticosteroids for over 14 days within 3 months prior to Screening or is likely to require treatment with systemic corticosteroids during the course of the study. Over the counter and prescription topical, inhaled, intranasal or injectable (for occasional use) corticosteroids are allowed.

Ages: 18 Years to 51 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 378 (Actual)
Dates: Start 2016-02-03 (Actual); Primary Completion 2018-02-14 (Actual); Study Completion 2019-01-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (105):
- United States (103):
  - Alabama Clinical Therapeutics, LLC /ID# 152258, Birmingham, Alabama
  - Choice Research, LLC /ID# 150988, Dothan, Alabama
  - Brown, Pearson, Guepet Gynecology /ID# 151020, Fairhope, Alabama
  - Mobile, Ob-Gyn, P.C. /ID# 144294, Mobile, Alabama
  - Mesa Obstetricians and Gynecol /ID# 149139, Mesa, Arizona
  - Visions Clinical Research-Tucs /ID# 151017, Tucson, Arizona
  - Core Healthcare Group /ID# 151016, Cerritos, California
  - Diagnamics Inc. /ID# 152469, Encinitas, California
  - HCP Clinical Research LLC /ID# 154434, Huntington Beach, California
  - Alliance Research Centers /ID# 149752, Laguna Hills, California
  - University of California, Los Angeles /ID# 149760, Los Angeles, California
  - Futura Research, Inc. /ID# 149759, Norwalk, California
  - Farid Yasharpour MD Medical Co /ID# 149770, San Fernando, California
  - Clinical Trial Investigators /ID# 152470, Tustin, California
  - Bayview Research Group LLC /ID# 153799, Valley Village, California
  - Emerson Clinical Research Inst /ID# 152348, Washington D.C., District of Columbia
  - Ideal Clinical Research Inc. /ID# 149757, Aventura, Florida
  - Seffner Premier Health Care, P /ID# 167480, Brandon, Florida
  - Olympian Clinical Research /ID# 149756, Clearwater, Florida
  - KO Clinical Research, LLC /ID# 144299, Fort Lauderdale, Florida
  - University of Florida /ID# 149751, Gainesville, Florida
  - Solutions Through Adv Rch /ID# 151021, Jacksonville, Florida
  - Meridien Research /ID# 167100, Kenneth City, Florida
  - Invictus Clinical Research Group,LLC /ID# 141859, Miami, Florida
  - Precision Research Org, LLC /ID# 144335, Miami Lakes, Florida
  - Suncoast Clinical Research /ID# 149765, New Port Richey, Florida
  - All Wmns HC of West Broward /ID# 144298, Plantation, Florida
  - Oncova Clinical Research, Inc. /ID# 149764, Saint Cloud, Florida
  - Physician Care Clin. Res., LLC /ID# 149766, Sarasota, Florida
  - Qps-Mra, Llc /Id# 144325, South Miami, Florida
  - Martin Health System Center /ID# 152263, Stuart, Florida
  - University of South Florida /ID# 149754, Tampa, Florida
  - Axcess Medical Research /ID# 149769, Wellington, Florida
  - Virtus Research Consultant,LLC /ID# 144296, Wellington, Florida
  - Paramount Research Solutions /ID# 149291, Alpharetta, Georgia
  - Agile Clinical Research Trials /ID# 167074, Atlanta, Georgia
  - Mount Vernon Clinical Res, LLC /ID# 144297, Atlanta, Georgia
  - Atlanta Women's Research Inst /ID# 144303, Atlanta, Georgia
  - Masters of Clinical Research, Inc. /ID# 167400, Augusta, Georgia
  - Georgia Regents University /ID# 144295, Augusta, Georgia
  - Meridian Clinical Research, LLC /ID# 149144, Savannah, Georgia
  - Gyn-Care, Inc. /ID# 149341, Smyrna, Georgia
  - Atlanta Gynecology Research Institute /ID# 151014, Suwanee, Georgia
  - Womens Healthcare Assoc, DBA /ID# 149762, Idaho Falls, Idaho
  - Advanced Clinical Research /ID# 149767, Meridian, Idaho
  - University of Chicago /ID# 152257, Chicago, Illinois
  - Affinity Clinical Research /ID# 167119, Oak Brook, Illinois
  - Center for Women's Research, Inc /ID# 144300, Palos Heights, Illinois
  - Women's Health Advantage /ID# 144301, Fort Wayne, Indiana
  - The Iowa Clinic /ID# 150105, West Des Moines, Iowa
  - PRN Professional Research Network of Kansas, LLC /ID# 152265, Wichita, Kansas
  - Bluegrass Clinical Research /ID# 150103, Louisville, Kentucky
  - Clinical Trials Management, LLC - Covington /ID# 144314, Covington, Louisiana
  - Women Under Study, LLC /ID# 144312, New Orleans, Louisiana
  - Baltimore Suburban Health /ID# 154638, Baltimore, Maryland
  - Womens Health Center /ID# 154209, Glen Burnie, Maryland
  - Maryland Ctr for Sexual Health /ID# 149778, Lutherville, Maryland
  - NECCR Fall River LLC /ID# 149584, Fall River, Massachusetts
  - Saginaw Valley Med Res Group /ID# 149768, Saginaw, Michigan
  - Accent Clinical Trials /ID# 149753, Las Vegas, Nevada
  - Jersey Shore University Medical Center /ID# 149779, Neptune City, New Jersey
  - Rowan University SOM /ID# 152697, Stratford, New Jersey
  - SUNY Downstate Medical Center /ID# 144311, Brooklyn, New York
  - Manhattan Medical Research /ID# 167077, New York, New York
  - Weill Cornell Medicine /ID# 149585, New York, New York
  - Montefiore Medical Center /ID# 149582, The Bronx, New York
  - Duplicate_Unified Women's Clinical Research-Fayetteville /ID# 149587, Fayetteville, North Carolina
  - Unified Women's Clinical Research-Greensboro /ID# 149588, Greensboro, North Carolina
  - Pinewest Ob-Gyn, Inc. /ID# 145671, High Point, North Carolina
  - Eastern Carolina Women's Centr /ID# 144309, New Bern, North Carolina
  - Wake Research Associates, LLC /ID# 144307, Raleigh, North Carolina
  - Clinical Inquest Center Ltd /ID# 148728, Beavercreek, Ohio
  - CTI Clinical Research Center /ID# 149761, Cincinnati, Ohio
  - The Christ Hospital /ID# 150104, Cincinnati, Ohio
  - Alpha Research Associates LLC /ID# 152471, Dayton, Ohio
  - Comprehensive Womens Care /ID# 144306, Westerville, Ohio
  - Family Medical Associates /ID# 145668, Levittown, Pennsylvania
  - University of Pennsylvania /ID# 149586, Philadelphia, Pennsylvania
  - Clinical Research of Philadelphia, LLC /ID# 151015, Philadelphia, Pennsylvania
  - Reading Hosp Clncl Trials Ofc /ID# 149583, West Reading, Pennsylvania
  - Holston Medical Group /ID# 149763, Bristol, Tennessee
  - Chattanooga Medical Research /ID# 145667, Chattanooga, Tennessee
  - Chattanooga Women for Women /ID# 167051, Hixson, Tennessee
  - The Jackson Clinic, PA /ID# 145670, Jackson, Tennessee
  - The Womens Physician Group /ID# 144317, Memphis, Tennessee
  - Access Clinical Trials, Inc. /ID# 167333, Nashville, Tennessee
  - Lotus Gynecology /ID# 149140, Austin, Texas
  - Inquest Clinical Research /ID# 149755, Baytown, Texas
  - Texas Health Presbyterian Hosp /ID# 149142, Dallas, Texas
  - Baylor College of Medicine /ID# 149141, Houston, Texas
  - The Woman's Hospital of Texas /ID# 144319, Houston, Texas
  - Centex Studies, Inc. - Houston /ID# 150106, Houston, Texas
  - BI Research Center /ID# 149143, Houston, Texas
  - FMC Science /ID# 151802, Lampasas, Texas
  - Willowbend Health and Wellness /ID# 144318, Plano, Texas
  - Clinical Trials of Texas,Inc. /ID# 144322, San Antonio, Texas
  - Center of Reproductive Medicin /ID# 167235, Webster, Texas
  - Southampton Women's Health /ID# 152325, Franklin, Virginia
  - Tidewater Physicians for Women /ID# 144321, Norfolk, Virginia
  - Clinical Research Partners, LLC /ID# 144310, Richmond, Virginia
  - Alliance Womens Health /ID# 152468, Richmond, Virginia
  - Zain Research /ID# 151018, Richland, Washington
  - Virginia Mason Medical Center /ID# 149758, Seattle, Washington
- Canada (2):
  - Medicor Research Inc. /ID# 153406, Greater Sudbury, Ontario
  - Victory Reproductive Care /ID# 150247, Windsor, Ontario

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Data requests can be submitted at any time and the data will be accessible for 12 months, with possible extensions considered.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information on the process, or to submit a request, visit the following link.
URL: https://www.abbvie.com/our-science/clinical-trials/clinical-trials-data-and-information-sharing/data-and-information-sharing-with-qualified-researchers.html

REFERENCES:
- [Derived] Simon JA, Stewart EA, Jewell S, Li M, Snabes MC. Impact of demographic and clinical factors on elagolix plus add-back therapy effects on patient-reported nonbleeding symptoms in women with heavy menstrual bleeding and uterine fibroids: a post hoc analysis of data from two clinical trials. F S Rep. 2024 Jun 14;5(3):285-295. doi: 10.1016/j.xfre.2024.06.002. eCollection 2024 Sep. PMID 39381651
- [Derived] Beck D, Winzenborg I, Liu M, Degner J, Mostafa NM, Noertersheuser P, Shebley M. Population Pharmacokinetics of Elagolix in Combination with Low-Dose Estradiol/Norethindrone Acetate in Women with Uterine Fibroids. Clin Pharmacokinet. 2022 Apr;61(4):577-587. doi: 10.1007/s40262-021-01096-w. Epub 2021 Dec 8. PMID 34878624
- [Derived] Stewart EA, Archer DF, Owens CD, Barnhart KT, Bradley LD, Feinberg EC, Gillispie-Bell V, Imudia AN, Liu R, Kim JH, Al-Hendy A. Reduction of Heavy Menstrual Bleeding in Women Not Designated as Responders to Elagolix Plus Add Back Therapy for Uterine Fibroids. J Womens Health (Larchmt). 2022 May;31(5):698-705. doi: 10.1089/jwh.2021.0152. Epub 2021 Sep 28. PMID 34582715
- [Derived] Muneyyirci-Delale O, Archer DF, Owens CD, Barnhart KT, Bradley LD, Feinberg E, Gillispie V, Hurtado S, Kim JH, Wang A, Wang H, Stewart EA. Efficacy and safety of elagolix with add-back therapy in women with uterine fibroids and coexisting adenomyosis. F S Rep. 2021 May 26;2(3):338-346. doi: 10.1016/j.xfre.2021.05.004. eCollection 2021 Sep. PMID 34553161
- [Derived] Beck D, Winzenborg I, Gao W, Mostafa NM, Noertersheuser P, Chiuve SE, Owens C, Shebley M. Integrating real-world data and modeling to project changes in femoral neck bone mineral density and fracture risk in premenopausal women. Clin Transl Sci. 2021 Jul;14(4):1452-1463. doi: 10.1111/cts.13006. Epub 2021 Apr 8. PMID 33650259
- [Derived] Schlaff WD, Ackerman RT, Al-Hendy A, Archer DF, Barnhart KT, Bradley LD, Carr BR, Feinberg EC, Hurtado SM, Kim J, Liu R, Mabey RG Jr, Owens CD, Poindexter A, Puscheck EE, Rodriguez-Ginorio H, Simon JA, Soliman AM, Stewart EA, Watts NB, Muneyyirci-Delale O. Elagolix for Heavy Menstrual Bleeding in Women with Uterine Fibroids. N Engl J Med. 2020 Jan 23;382(4):328-340. doi: 10.1056/NEJMoa1904351. PMID 31971678

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Eligible participants were randomized in a 1:1:2 ratio to 1 of 3 treatment groups: placebo, elagolix 300 mg BID, or elagolix 300 mg twice daily (BID) plus estradiol/norethindrone acetate (E2/NETA) once daily (QD).
Groups:
- Placebo: Placebo for both elagolix BID and E2/NETA QD
Period: Treatment Period
Arm/Group | Placebo | Elagolix | Elagolix + E2/NETA
Started (randomized and treated) | 94 | 95 | 189
Completed | 72 (completed treatment period) | 69 (completed treatment period) | 148 (completed treatment period)
Not Completed | 22 | 26 | 41
Period: Post-Treatment Follow-Up Period
Arm/Group | Placebo | Elagolix | Elagolix + E2/NETA
Started | 14 | 25 | 59
Completed | 9 | 18 | 42
Not Completed | 5 | 7 | 17
Not completed — Withdrawal by Subject | 1 | 2 | 8
Not completed — Lost to Follow-up | 2 | 3 | 4
Not completed — Other | 2 | 1 | 1
Not completed — Required Surgery/Invasive Intervention | 0 | 0 | 3
Not completed — Non-Compliance | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Elagolix | Elagolix + E2/NETA | Total
Number analyzed (Participants) | 94 | 95 | 189 | 378
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.5 (5.43) | 42.2 (5.41) | 42.5 (5.33) | 42.4 (5.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94 | 95 | 189 | 378
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 17 | 31 | 59
  Not Hispanic or Latino | 83 | 78 | 158 | 319
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 2 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 2 | 2
  Black or African American | 63 | 66 | 124 | 253
  White | 30 | 27 | 59 | 116
  More than one race | 0 | 0 | 3 | 3
  Unknown or Not Reported | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Meeting the Criteria for Responder
Description: Percentage of responders, defined as participants who met the following conditions:
  * Menstrual blood loss (MBL) volume < 80 mL during the Final Month (the last 28 days prior to and including the Reference Day, which is defined as the last visit date during the Treatment Period (last treatment visit date) or the last dose date if there are evaluable alkaline hematin data after the last treatment visit date and prior to or on the last dose date), and
  * ≥ 50% reduction in MBL volume from Baseline to the Final Month.
  Participants who prematurely discontinued study drug due to "lack of efficacy," "requires surgery or invasive intervention for treatment of uterine fibroids," or "adverse events" were considered non-responders regardless of whether she meets the two aforementioned responder criteria or not.
Time Frame: Final Month (the last 28 days prior to and including the Reference Day), up to Month 6
Population: All randomized and treated participants.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Elagolix | Elagolix + E2/NETA
Number analyzed (Participants) | 94 | 95 | 189
percentage of participants | 10.5 | 76.9 | 76.5
Statistical Analysis 1: Comparison: Placebo vs Elagolix; Test type: Superiority; p < 0.001, Regression, Logistic — The P value for test of difference is by pooling the results from a logistic regression model including treatment as the main effect and baseline MBL volume as a covariate in each data set from multiple imputation; Odds Ratio (OR) = 28.73, 95% CI 2-sided [12.248 to 67.387]
Statistical Analysis 2: Comparison: Placebo vs Elagolix + E2/NETA; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 28.31, 95% CI 2-sided [13.042 to 61.431]

2. Secondary Outcome: Change From Baseline in MBL Volume to the Final Month
Description: Baseline MBL volume was defined as the mean of total MBL volume from all the qualified menstrual cycles during the Screening Period, in which the total MBL volume is from all validated and non-validated sanitary products and the MBL volume of validated sanitary products only (excluding non-validated sanitary products) was greater than 80 mL.
  The Reference Day is defined as the last visit date during the Treatment Period (last treatment visit date) or the last dose date if there are evaluable alkaline hematin data after the last treatment visit date and prior to or on the last dose date.
Time Frame: Baseline and Final Month (the last 28 days prior to and including the Reference Day), up to Month 6
Population: All randomized and treated participants.
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Placebo | Elagolix | Elagolix + E2/NETA
Number analyzed (Participants) | 94 | 95 | 189
mL | -4.3 (15.44) | -198.8 (15.44) | -168.8 (10.72)
Statistical Analysis 1: Comparison: Placebo vs Elagolix; Test type: Superiority; p < 0.001, ANCOVA — The P value for test of difference between each elagolix treatment group and placebo is by pooling the results from an ANCOVA model with treatment as the main effect and baseline MBL volume as a covariate in each dataset from multiple imputation; LS Mean of Difference = -194.5, Standard Error of Mean 21.70
Statistical Analysis 2: Comparison: Placebo vs Elagolix + E2/NETA; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean of Difference = -164.6, Standard Error of Mean 18.87

3. Secondary Outcome: Percentage of Participants With Suppression of Bleeding at the Final Month
Description: Suppression of bleeding is defined as having 0 days of bleeding (spotting is allowed) during the Final Month with the interval starting from Study Day 11.
  The Reference Day is defined as the last visit date during the Treatment Period (last treatment visit date) or the last dose date if there are evaluable alkaline hematin data after the last treatment visit date and prior to or on the last dose date.
Time Frame: Final Month (the last 28 days prior to and including the Reference Day), up to Month 6
Population: All randomized and treated participants with an assessment
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Elagolix | Elagolix + E2/NETA
Number analyzed (Participants) | 85 | 81 | 172
percentage of participants | 4.7 | 88.9 | 61.0
Statistical Analysis 1: Comparison: Placebo vs Elagolix; Test type: Superiority; p < 0.001, chi-square or Fisher's exact test — The P value is calculated based on chi-square test (or Fisher's exact test if ≥ 20% of the cells have expected cell count < 5); Between-Group Difference (%) = 84.2, 95% CI 2-sided [75.99 to 92.37]
Statistical Analysis 2: Comparison: Placebo vs Elagolix + E2/NETA; Test type: Superiority; p < 0.001, chi-square or Fisher's exact test — [p-value comment as in outcome 3, analysis 1]; Between-Group Difference (%) = 56.3, 95% CI 2-sided [47.77 to 64.91]

4. Secondary Outcome: Change From Baseline in MBL Volume to Month 6
Description: Baseline MBL volume was defined as the mean of total MBL volume from all the qualified menstrual cycles during the Screening Period, in which the total MBL volume is from all validated and non-validated sanitary products and the MBL volume of validated sanitary products only (excluding non-validated sanitary products) was greater than 80 mL.
Time Frame: Month 0 (Baseline), Month 6
Population: All randomized and treated participants with an assessment at given time point.
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Placebo | Elagolix | Elagolix + E2/NETA
Number analyzed (Participants) | 64 | 53 | 124
mL | 28.5 (16.68) | -223.7 (17.98) | -198.1 (11.89)
Statistical Analysis 1: Comparison: Placebo vs Elagolix; Test type: Superiority; p < 0.001, mixed model repeated measures — The P value is from mixed models repeated measures (MMRM) with treatment, month, and an interaction between treatment and month as fixed effect factors, and baseline MBL volume as a covariate comparing each elagolix treatment group with placebo; LS Mean of Difference = -252.3, Standard Error of Mean 24.53
Statistical Analysis 2: Comparison: Placebo vs Elagolix + E2/NETA; Test type: Superiority; p < 0.001, mixed model repeated measures — [p-value comment as in outcome 4, analysis 1]; LS Mean of Difference = -226.6, Standard Error of Mean 20.50

5. Secondary Outcome: Change From Baseline in MBL Volume to Month 3
Description: as for outcome 4
Time Frame: Month 0 (Baseline), Month 3
Population: All randomized and treated participants with an assessment at given time point.
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Placebo | Elagolix | Elagolix + E2/NETA
Number analyzed (Participants) | 78 | 72 | 157
mL | -14.2 (11.57) | -211.1 (11.96) | -200.3 (8.17)
Statistical Analysis 1: Comparison: Placebo vs Elagolix; Test type: Superiority; p < 0.001, mixed model repeated measures — The P value is from MMRM with treatment, month, and an interaction between treatment and month as fixed effect factors, and baseline MBL volume as a covariate comparing each elagolix treatment group with placebo; LS Mean of Difference = -196.9, Standard Error of Mean 16.66
Statistical Analysis 2: Comparison: Placebo vs Elagolix + E2/NETA; Test type: Superiority; p < 0.001, mixed model repeated measures — [p-value comment as in outcome 5, analysis 1]; LS Mean of Difference = -186.1, Standard Error of Mean 14.18

6. Secondary Outcome: Percentage of Participants With Baseline Hemoglobin <= 10.5 g/dL Who Have an Increase in Hemoglobin > 2 g/dL at Month 6
Time Frame: Month 0 (Baseline), Month 6
Population: All randomized and treated participants with baseline hemoglobin <= 10.5 g/dL and an assessment at Month 6.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Elagolix | Elagolix + E2/NETA
Number analyzed (Participants) | 24 | 25 | 48
percentage of participants | 20.8 | 40.0 | 50.0
Statistical Analysis 1: Comparison: Placebo vs Elagolix; Test type: Superiority; p = 0.146, chi-square or Fisher's exact test — [p-value comment as in outcome 3, analysis 1]; Between-Group Difference (%) = 19.2, 95% CI 2-sided [-5.99 to 44.32]
Statistical Analysis 2: Comparison: Placebo vs Elagolix + E2/NETA; Test type: Superiority; p = 0.017, chi-square or Fisher's exact test — [p-value comment as in outcome 3, analysis 1]; Between-Group Difference (%) = 29.2, 95% CI 2-sided [7.62 to 50.71]

7. Secondary Outcome: Change From Baseline in MBL Volume to Month 1
Description: as for outcome 4
Time Frame: Month 0 (Baseline), Month 1
Population: All randomized and treated participants with an assessment at given time point.
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Placebo | Elagolix | Elagolix + E2/NETA
Number analyzed (Participants) | 88 | 83 | 175
mL | -2.1 (14.31) | -196.6 (14.74) | -127.0 (10.14)
Statistical Analysis 1: Comparison: Placebo vs Elagolix; Test type: Superiority; p < 0.001, mixed model repeated measures — [p-value comment as in outcome 5, analysis 1]; LS Mean of Difference = -194.5, Standard Error of Mean 20.56
Statistical Analysis 2: Comparison: Placebo vs Elagolix + E2/NETA; Test type: Superiority; p < 0.001, mixed model repeated measures — [p-value comment as in outcome 5, analysis 1]; LS Mean of Difference = -125.0, Standard Error of Mean 17.55

ADVERSE EVENTS:
Time Frame: From first dose of study drug through 6 months of treatment with a 30-day follow-up period for participants who did not enroll in the extension study (Study M12-816). Mean (SD) treatment exposure was 160.3 (51.75), 155.2 (65.19), and 158.7 (54.68) days for the Placebo, Elagolix, and Elagolix and E2-NETA arms, respectively
Description: Treatment-emergent adverse events are presented.
Groups:
- Elagolix + E2-NETA: Elagolix 300 mg BID and E2/NETA (estradiol 1.0 mg/norethindrone acetate 0.5 mg) QD
Arm/Group | Placebo | Elagolix | Elagolix + E2-NETA
All-Cause Mortality (participants affected / at risk) | 0/94 | 0/95 | 0/189
Serious Adverse Events (participants affected / at risk) | 1/94 | 4/95 | 7/189
Other Adverse Events (participants affected / at risk) | 34/94 | 58/95 | 80/189
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=94) | Elagolix (N=95) | Elagolix + E2-NETA (N=189)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
HYPERTHYROIDISM (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
CHOLELITHIASIS (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1)
APPENDICITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
CELLULITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OBESITY (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
ABORTION COMPLETE (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0)
ANXIETY (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
DYSFUNCTIONAL UTERINE BLEEDING (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
DYSMENORRHOEA (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
MENORRHAGIA (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
PELVIC PAIN (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=94) | Elagolix (N=95) | Elagolix + E2-NETA (N=189)
NAUSEA (Gastrointestinal disorders) | 9 (11) | 4 (4) | 14 (15)
FATIGUE (General disorders) | 5 (5) | 3 (3) | 10 (10)
NASOPHARYNGITIS (Infections and infestations) | 8 (9) | 4 (4) | 10 (11)
URINARY TRACT INFECTION (Infections and infestations) | 5 (6) | 2 (2) | 12 (12)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (5) | 9 (10)
HEADACHE (Nervous system disorders) | 5 (6) | 13 (14) | 20 (21)
LIBIDO DECREASED (Psychiatric disorders) | 2 (2) | 3 (3) | 10 (10)
MOOD SWINGS (Psychiatric disorders) | 2 (2) | 6 (6) | 6 (8)
DYSMENORRHOEA (Reproductive system and breast disorders) | 6 (6) | 0 (0) | 6 (6)
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 5 (6) | 24 (24) | 20 (21)
HOT FLUSH (Vascular disorders) | 4 (4) | 41 (41) | 37 (37)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2017-10-06): https://cdn.clinicaltrials.gov/large-docs/94/NCT02691494/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-02): https://cdn.clinicaltrials.gov/large-docs/94/NCT02691494/SAP_001.pdf